CLINICAL TRIAL: NCT02054325
Title: A Randomized Triple-blind Study Protocol Comparing Polidocanol Versus Hypertonic Glucose for Sclerotherapy in Treatment of Reticular Veins at the Lower Limbs.
Brief Title: Study Protocol Comparing Polidocanol Versus Hypertonic Glucose for Treatment of Reticular Veins
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: UPECLIN HC FM Botucatu Unesp (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Dr Matheus Bertanha, Professor, UPECLIN HC FM Botucatu Unesp
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CEP 4127.2012
Record Dates: First submitted 2014-02-01; First posted 2014-02-04 (Estimated); Results first posted 2017-01-27 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2016-11

CONDITIONS: Varicose Veins
Keywords: Sclerotherapy; varicose veins; veins
MeSH Terms: conditions — Varicose Veins | interventions — Polidocanol; Glucose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Polidocanol with Glucose (Active Comparator): An application session 0.2% Polidocanol + 70% Glucose to treat reticular veins of the lower limb selected, with a maximum volume of 5 ml.
  Interventions: Drug: Polidocanol with Glucose
- Glucose (Active Comparator): An application session 75% Glucose to treat reticular veins of the lower limb selected, with a maximum volume of 5ml.
  Interventions: Drug: Glucose

INTERVENTIONS:
Drug: Polidocanol with Glucose — An application session 0.2% Polidocanol + 70% Glucose to treat reticular veins of the lower limb selected, with a maximum volume of 5 ml. Return to a week to investigate the adverse effects and 2 months for proof of efficacy and adverse effects
  Other Names: Dodecylpolyethyleneglycolether; Aethoxysklerol; Varithena
  Arms: Polidocanol with Glucose
Drug: Glucose — An application session 75% Glucose to treat reticular veins of the lower limb selected, with a maximum volume of 5 ml. Return to a week to investigate the adverse effects and 2 months for proof of efficacy and adverse effects
  Other Names: Dextrose
  Arms: Glucose

SUMMARY:
It will be done a randomized triple-blind study comparing 0,2% polidocanol versus 75% hypertonic glucose of sclerotherapy in lower limbs´ reticular veins. It will be included only adult women with reticular veins on the side of the thighs and mild venous insufficiency (CEAP 1). The primary endpoint will be efficacy, and secondary will be safety.

DETAILED DESCRIPTION:
Background. The prevalence of chronic venous disease is high in the general population, mainly in young women, and in milder cases the usual complaint is aesthetic. Various techniques are used for treatment of mild varicose disease, including surgical treatment, laser ablation and sclerotherapy. Reticular veins are those with less than 3mm diameter, bluish and important contribution to the aesthetic damage, and sometimes they are related to local pain and recurrence after treatment of telangiectasias. There is no consensus in the literature about the effectiveness of treatment with sclerotherapy, despite of being an usual procedure with different chemicals.

Methods and design. One hundred lower limbs of healthy women between 18 and 69 years will be triple blind randomized to receive treatment with polidocanol 0.2% diluted in 70% hypertonic glucose versus 75% hypertonic glucose for sclerotherapy treatment of reticular veins. The patients will be examined and clinically classified. It will be included patients with reticular veins sited at out's thigh/leg, measuring at least 10cm long, and only one extremity will be included per patient. The patients with varicose disease CEAP 2 or more will not be included. The treatment will be carried out in only one session and the medication volume not exceeding 5 ml. Clinical follow-up protocols will be filled on regular visits on days 0 - 7 - 60 concomitantly with photograph documentation. Supplementary examination for venous mapping with ultrasound pretreatment is performed for all patients.

Discussion. This prospective controlled double-blind randomized trial aims to verify and compare the efficacy and safety for sclerotherapy treatment of reticular veins of the lower limbs. The results may help physicians to choose the best sclerotherapy treatment for reticular veins.

ELIGIBILITY:
Inclusion Criteria:

* females
* with at least 10 cm from the lateral reticular veins of the leg or thigh of the leg
* clinical classification of chronic venous disease C1(mild venous disease),
* minimum age of 18 year-old and maximum age 69 year-old
* agreement with the study
* signing the free and informed consent ( IC)
* not use anticoagulant drugs .

Exclusion Criteria:

* male
* varicose disease in any quantity or location with clinical classification of chronic venous disease different of C1(mild venous disease)
* restrict mobility
* arterial insufficiency
* be allergic to any substance that may be related to the study drugs
* any cause of dermatitis on application site
* free of comorbidities clinically serious as diabetes mellitus, heart failure, respiratory failure, uncontrolled hypertension with medication, and uncontrolled hypothyroidism
* pregnancy
* previous deep vein thrombosis (DVT)
* family history of DVT
* thrombophilia
* do not agree with the search terms

Ages: 18 Years to 69 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2012-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matheus Bertanha, Professor, Principal Investigator — UPECLIN HC FM Botucatu Unesp
Locations (1):
- School of Medicine at Botucatu- Paulista State University- UNESP, São Paulo, Brazil, Botucatu, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided
We intend to present data when publish the original article.

REFERENCES:
- [Derived] Bertanha M, Jaldin RG, Moura R, Pimenta REF, Mariuba JVO, Lucio Filho CEP, Alcantara GP, Padovani CR, Yoshida WB, Sobreira ML. Sclerotherapy for Reticular Veins in the Lower Limbs: A Triple-Blind Randomized Clinical Trial. JAMA Dermatol. 2017 Dec 1;153(12):1249-1255. doi: 10.1001/jamadermatol.2017.3426. PMID 28973414
- [Derived] Bertanha M, Sobreira ML, Pinheiro Lucio Filho CE, de Oliveira Mariuba JV, Farres Pimenta RE, Jaldin RG, Moroz A, Moura R, Rollo HA, Yoshida WB. Polidocanol versus hypertonic glucose for sclerotherapy treatment of reticular veins of the lower limbs: study protocol for a randomized controlled trial. Trials. 2014 Dec 19;15:497. doi: 10.1186/1745-6215-15-497. PMID 25527165

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Some patients (n=6) were withdrawn because did not appear at the previous scheduled appointments, and were replaced for new ones. In order to avoid loss of individuals we have decided to include 6 more patients.
Period: Overall Study
Arm/Group | Polidocanol With Glucose | Glucose
Started | 51 | 55
Completed | 43 | 50
Not Completed | 8 | 5
Not completed — Lost to Follow-up | 8 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Polidocanol With Glucose | Glucose | Total
Number analyzed (Participants) | 43 | 50 | 93
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 43 | 50 | 93
  >=65 years | 0 | 0 | 0
Gender [Count of Participants; unit: Participants]
  Female | 43 | 50 | 93
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Efficacy in Treating Reticular Veins by Photographs: Mean Percent Reticular Vein Disappearance Two Months After Treatment.
Description: Photographs were performed pretreatment and two months after the treatment, these were analyzed for efficacy in treat reticular veins by two blind analyzers objectively with measurement through the use of free software ImageJ.
Time Frame: Mean Percent of reticular vein disappearance two months after treatment
Measure: Mean (Standard Deviation); unit: % of Reticular Veins that Disappeared
Arm/Group | Polidocanol With Glucose | Glucose
Number analyzed (Participants) | 43 | 50
% of Reticular Veins that Disappeared | 95.17 (9.09) | 85.40 (17.04)

2. Secondary Outcome: The Safety of the Treatment: Mean Percent of Skin Hyperpigmentation Two Months After Treatment
Description: Skin hyperpigmentation was defined as a brownish hue stain superimposing the previous treated vein site (by visual photographic analyses). Skin hyperpigmentation was firstly evaluated according to its occurence and labeled as "Yes" or "No". Afterwards, when there was stain in the previous treated area, a line was drawn on the stain with Image J software , and the Mean Percent of Skin Hyperpigmentation was proportionaly compared with length of vein treated, previuos mesuread (mean and SD).
Time Frame: Two months after treatment.
Measure: Mean (Standard Deviation); unit: Percent of Skin Hyperpigmentation
Arm/Group | Polidocanol With Glucose | Glucose
Number analyzed (Participants) | 43 | 50
Percent of Skin Hyperpigmentation | 5.75 (7.02) | 9.66 (11.67)

ADVERSE EVENTS:
Time Frame: Right after two months post procedure
Description: Hyperpigmentation: Linear measure above the projection area of hyperpigmentation post procedure. The length of this line was provided by the Image J software (ImageJ is a public domain, Java-based image processing program developed at the National Institutes of Health)
Arm/Group | Polidocanol With Glucose | Glucose
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/50
Other Adverse Events (participants affected / at risk) | 22/43 | 31/50
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Polidocanol With Glucose (N=43) | Glucose (N=50)
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 22 | 31 — Dark pigmentation of skin after injection

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes